CLINICAL TRIAL: NCT00001754
Title: Clinical and Molecular Manifestations of Human Skeletal Dysplasias and Short Stature
Brief Title: Study of Skeletal Disorders and Short Stature
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 980119; 98-HG-0119
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-06

CONDITIONS: Developmental Bone Disease; Dwarfism; Skeletal Dysplasias
Keywords: Dwarfism; Gene Mapping; Linkage; Mutation Analysis; Skeletal Biology; Brachydactyly Types C & E; Cartilage-Hair Hypoplasia; Ellis Van Crevald; FgFR-3; Proximal Symphalangism; Pyknodysotosis; Schmid Metaphyseal; Short Stature; Skeletal Dysplasia; Type II Collagen Disorder
MeSH Terms: conditions — Bone Diseases, Developmental; Dwarfism; Cartilage-hair hypoplasia; Cushing's symphalangism; Mucopolysaccharidosis IV

SUMMARY:
This study will determine the genes responsible for skeletal dysplasias (disorders of the skeleton) and short stature and define the range and type of medical problems they cause over time. It will investigate whether specific gene changes cause specific medical problems in these disorders and identify the signs and symptoms upon which their diagnoses must be based.

Individuals with short stature or with a skeletal dysplasia known or suspected to be caused by a gene mutation (change) may be eligible for this study. Family members may also participate. Skeletal dysplasias under study include: achondroplasia, hypochondroplasia, achondrogenesis type II, hypochondrogenesis, Kniest dysplasia, spondyloepiphyseal dysplasias, Stickler syndrome; Shmid and Jansen metaphyseal dysplasias; pyknodysotosis, proximal symphalangism, brachydactyly types B C and E, Ellis van Creveld and related disorders, metatrophic chondrodysplasias, cartilage-hair hypoplasia and disorders with a skeletal abnormality that have not yet been defined but might be the result of a genetic defect.

Patients will talk with two genetics specialists who will explain the study and its possible implications for the patient and family and answer questions. The patient's medical records will be reviewed, a personal and family history will be taken, and a physical examination will be done. Various other procedures that may be done include drawing up to 6 tablespoons of blood, some of which will be used for DNA (genetic) studies, X-rays, echocardiography (ultrasound of the heart), magnetic resonance imaging (MRI), eye examination, hearing test, sleep study, sperm analysis and skin biopsy (surgical removal of a small piece of skin done under local anesthetic). There may be additional evaluations by specialists in rheumatology, rehabilitation medicine and orthopedics. When the tests and examinations are completed (after 2 to 3 days), a doctor will discuss the results with the patient. Patients whose DNA studies show that a gene change is responsible for their disorder will meet with a genetics nurse or counselor to review the results, express their feelings and ask any questions they may have. Patients may be asked to return to NIH every 6 months to 2 years for continued follow-up. Medical management will be provided primarily by the patient's own physician.

Participating family members will be interviewed by telephone about their personal and family health history and will have a blood sample drawn for DNA testing. If a gene change is found that is responsible for the bone disorder or growth problem in the family, arrangements will be made for the family member to discuss the implications of the findings with a genetics specialist.

DETAILED DESCRIPTION:
We will investigate the clinical manifestations and molecular genetic defects of human skeletal dysplasias and generalized short stature. Families with skeletal dysplasias or short stature of known or suspected genetic basis will be enrolled. Affected individuals or individuals suspected of having a skeletal dysplasia will undergo periodic clinical assessment and genetic analyses for the purpose of: 1) definition and characterization of phenotype, 2) determination of the natural history of the disorder, and 3) genotype/phenotype correlation. Genetic linkage studies may be performed for disorders in which the genetic bases is not yet known.

ELIGIBILITY:
Patients with known or suspected skeletal dysplasias or short stature and their family members of any age will be recruited worldwide from diverse medical communities including genetics, orthopedics, ophthalmology, and pediatrics.

DISEASE CATEGORY I:

Individuals and family members with a suspected or an established diagnosis of any FGFR3 disorder, type II collagen disorder, Schmid metaphyseal dysplasia, pyknodysostosis, proximal symphalangism, or brachydactyly type C.

DISEASE CATEGORY II:

Individuals and family members with a suspected or an established diagnosis of a skeletal dysplasia in which the disease gene is not yet known, including: Ellis van Crevald, brachydactyly types B and E, and cartilage-hair hypoplasia.

DISEASE CATEGORY III:

Individuals and family members who have previously uncharacterized systemic manifestations suggestive of a skeletal dysplasias, with clinical findings of: disproportionate or proportionate short stature; and/or cleft palate; and/or detached retina; and/or history of loose joints or frequent joint dislocation; and/or history of, or family history of, premature arthritis.

Short Stature Category I: Individuals with generalized short stature and their family members. This includes adults with abnormal stature as statistically defined from standardized growth charts.

Must be able to give informed consent, older children (greater than or equal to 7 years old) who do not give assent, or persons who are wards of the state will be excluded from the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600
Dates: Start 1998-06; Study Completion 2001-05

CONTACTS AND LOCATIONS:
Locations (1):
- National Human Genome Research Institute (NHGRI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Bellus GA, Hefferon TW, Ortiz de Luna RI, Hecht JT, Horton WA, Machado M, Kaitila I, McIntosh I, Francomano CA. Achondroplasia is defined by recurrent G380R mutations of FGFR3. Am J Hum Genet. 1995 Feb;56(2):368-73. PMID 7847369
- [Background] Bellus GA, McIntosh I, Smith EA, Aylsworth AS, Kaitila I, Horton WA, Greenhaw GA, Hecht JT, Francomano CA. A recurrent mutation in the tyrosine kinase domain of fibroblast growth factor receptor 3 causes hypochondroplasia. Nat Genet. 1995 Jul;10(3):357-9. doi: 10.1038/ng0795-357. PMID 7670477
- [Background] Bogaert R, Tiller GE, Weis MA, Gruber HE, Rimoin DL, Cohn DH, Eyre DR. An amino acid substitution (Gly853-->Glu) in the collagen alpha 1(II) chain produces hypochondrogenesis. J Biol Chem. 1992 Nov 5;267(31):22522-6. PMID 1429602